CLINICAL TRIAL: NCT06890520
Title: Neurometabolic Profile of Individuals With Primary Mitochondrial Disease
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 24-022407
Record Dates: First submitted 2025-02-19; First posted 2025-03-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Primary Mitochondrial Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Genetically Confirmed Primary Mitochondrial Disease: Individuals with Genetically Confirmed Primary Mitochondrial Disease
- Healthy Controls: Individuals who have no history of Primary Mitochondrial Disease

SUMMARY:
Primary Mitochondrial Disease (PMD) is a genetic neurometabolic disorder, leading to central nervous system degeneration and increased risk of early mortality. There is a strong link between the pathophysiology of mitochondrial disease and biomarkers related to the biochemistry of redox imbalance, involving the levels of glutathione. Investigators will use Magnetic Resonance Imaging and Spectroscopy to non-invasively measure glutathione and other chemicals in the brain to identify redox imbalance in patients with PMD.

DETAILED DESCRIPTION:
Primary Mitochondrial Disease (PMD) is a genetic neurometabolic disorder, leading to the degeneration of the central nervous system (CNS) and increased risk of early mortality. PMD can be caused by mutations in several genes in the mitochondrial DNA as well as nuclear DNA. Although a rare disease, PMD can significantly impact quality of life, increasing healthcare costs and caregiver burden. There is a lack of non-invasive, validated, and objective markers of mitochondrial function. However, there is a strong link between the pathophysiology of mitochondrial disease and biomarkers related to the biochemistry of redox imbalance, involving the levels of glutathione (GSH). Redox imbalance can also result in the overgeneration of radicals, causing neuronal damage. With the advancement in magnetic resonance techniques, the investigators can measure the levels of GSH and other neurochemicals non-invasively in the brain. Investigators in this proposal will use Magnetic Resonance Spectroscopy and Imaging (MRS and MRI) to measure brain chemicals, structure, and function.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 8 and 75 years, inclusive
* Genetically confirmed primary mitochondrial disease
* Receiving standard-of-care treatment including mitochondrial supplements that may include N-acetylcysteine (NAC), a precursor of glutathione

Inclusion Criteria for Healthy Controls:

* Must be between 8 and 75 years, inclusive

Exclusion Criteria:

* MRI contraindications
* In the investigator's opinion, inability to fully comply with research procedures
* Active self-reported alcohol and/or substance abuse, including tobacco-use
* A pacemaker; any metal-based medical or non-medical devices/implants; any non-removable metal-based object (e.g., body piercings, jewelry, etc.) that cannot be cleared through radiologic evaluation
* Any history of intraocular injury or fragment in or around the orbit that cannot be cleared through radiologic evaluation
* Any history of bullet, shrapnel, or stabbing wounds that cannot be cleared through radiologic evaluation
* Past or current employment involving (or exposure to) a metal grinder (e.g., at a construction worksite)
* At the discretion of the principal investigator (PI), any medical condition that will interfere with or prevent the safe completion of the study
* Any female participant with childbearing potential who is knowingly pregnant or suspects that she is pregnant will be removed from the study. (Although there are no known risks of MRI on pregnant females or fetuses, there is a possibility of yet undiscovered pregnancy-related risks. Since there is no direct benefit from participating in this protocol for pregnant females, they will be excluded to ensure their long-term safety and that of their unborn fetus.)
* To note, for this protocol, participants are instructed to lie still in the MRI scanner; there is no contrast or sedation. Participants who do not possess the cognitive and / or physical abilities to perform these procedures will not be included.

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is an observational study among two study population groups: genetically confirmed PMD patients and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Assess group differences in brain chemical levels in Genetically Confirmed Primary Mitochondrial Disease (GC-PMD) compared to healthy controls (HC) | Approximately 1 day
  Metabolite concentrations from H Magnetic Resonance Spectroscopy (MRS) will be processed in Osprey followed by linear combination modelling of MRS spectra. Water-scaled metabolite estimates will be calculated and corrected for tissue composition and relaxation effects to generate metabolite concentrations.

SECONDARY OUTCOMES:
Change in Plasma glutathione levels in Genetically Confirmed Primary Mitochondrial Disease (GC-PMD) compared to healthy controls (HC) | Approximately 1 day
  Analyze and report plasma glutathione levels (µM) in affected cases versus healthy controls. Glutathione is an antioxidant that protects cells from oxidative stress and detoxification. Differences between the two groups is anticipated.
Change in Corticol Thickness in Genetically Confirmed Primary Mitochondrial Disease (GC-PMD) compared to healthy controls (HC) | Approximately 1 day
  Morphometric analyses and reporting of cortical thickness, surface area, and volume in affected cases versus healthy controls. Reporting cortical thickness involves using structural magnetic resonance imaging (MRI) to measure the width of the gray matter of the cortex, typically in millimeters, and analyzing regional variations to asses brain structure and function.
Change in Cerebral Blood Flow in Genetically Confirmed Primary Mitochondrial Disease (GC-PMD) compared to healthy controls (HC) | Approximately 1 day
  Cerebral blood flow imaging (using spin labeling or similar), analyses, and reporting in affected cases versus healthy controls. Studying blood flow in the brain can assess for cerebrovascular disease.

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided